CLINICAL TRIAL: NCT01545934
Title: Preventing Excessive Gestational Weight Gain in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Suzanne Phelan, Principle Investigator, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U01 HL114377A; U01HL114377 (NIH)
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Obesity
Keywords: Overweight; Obese; Pregnancy; Weight Gain
MeSH Terms: conditions — Obesity; Overweight; Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention)
- Lifestyle intervention (Experimental)
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — The intervention is a multicomponent program designed to prevent excessive gestational weight gain in obese women through modifications of diet, exercise, and behavioral strategies during pregnancy.
  Arms: Lifestyle intervention

SUMMARY:
The purpose of this study is to study the effects of a multicomponent lifestyle intervention that includes partial meal replacements as a means to prevent excessive gestational weight gain in obese women. The primary hypothesis is that the intervention will reduce the rate of gestational weight gain compared with standard care.

ELIGIBILITY:
Inclusion criteria:

* Over 18 years old
* < 16 weeks gestation
* BMI >= 25
* Willing to consent

Exclusion Criteria:

* Pregnant with Twins
* Untreated medical or psychological problem
* Inability to be physically active

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD, Principal Investigator — Cal Poly
Locations (2):
- United States (2):
  - California Polytechnic State University, San Luis Obispo, California
  - Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Cabre HE, Drews KL, Pomeroy J, Keadle SK, Arteaga SS, Franks PW, Haire-Joshu D, Knowler WC, Pi-Sunyer X, Van Horn L, Wing RR, Cahill AG, Clifton RG, Couch KA, Gallager D, Josefson JL, Joshipura K, Klein S, Martin CK, Peaceman AM, Phelan S, Thom EA, Redman LM; LIFE-Moms Research Group. LIFE-Moms: effects of multicomponent lifestyle randomized control trial on physical activity during pregnancy in women with overweight and obesity. Int J Behav Nutr Phys Act. 2025 Sep 30;22(1):119. doi: 10.1186/s12966-025-01805-9. PMID 41029405
- [Derived] Flanagan EW, Drews KL, Cade WT, Franks PW, Gallagher D, Phelan S, Van Horn L, Redman LM. Metabolic Health and Heterogenous Outcomes of Prenatal Interventions: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2528264. doi: 10.1001/jamanetworkopen.2025.28264. PMID 40839263
- [Derived] Redman LM, Drews KL, Klein S, Horn LV, Wing RR, Pi-Sunyer X, Evans M, Joshipura K, Arteaga SS, Cahill AG, Clifton RG, Couch KA, Franks PW, Gallagher D, Haire-Joshu D, Martin CK, Peaceman AM, Phelan S, Thom EA, Yanovski SZ, Knowler WC; LIFE-Moms Research Group. Attenuated early pregnancy weight gain by prenatal lifestyle interventions does not prevent gestational diabetes in the LIFE-Moms consortium. Diabetes Res Clin Pract. 2021 Jan;171:108549. doi: 10.1016/j.diabres.2020.108549. Epub 2020 Nov 22. PMID 33238176
- [Derived] Phelan S, Wing RR, Brannen A, McHugh A, Hagobian T, Schaffner A, Jelalian E, Hart CN, Scholl TO, Munoz-Christian K, Yin E, Phipps MG, Keadle S, Abrams B. Does Partial Meal Replacement During Pregnancy Reduce 12-Month Postpartum Weight Retention? Obesity (Silver Spring). 2019 Feb;27(2):226-236. doi: 10.1002/oby.22361. Epub 2018 Nov 13. PMID 30421864
- [Derived] Peaceman AM, Clifton RG, Phelan S, Gallagher D, Evans M, Redman LM, Knowler WC, Joshipura K, Haire-Joshu D, Yanovski SZ, Couch KA, Drews KL, Franks PW, Klein S, Martin CK, Pi-Sunyer X, Thom EA, Van Horn L, Wing RR, Cahill AG; LIFE-Moms Research Group. Lifestyle Interventions Limit Gestational Weight Gain in Women with Overweight or Obesity: LIFE-Moms Prospective Meta-Analysis. Obesity (Silver Spring). 2018 Sep;26(9):1396-1404. doi: 10.1002/oby.22250. Epub 2018 Sep 6. PMID 30230252
- [Derived] Phelan S, Wing RR, Brannen A, McHugh A, Hagobian TA, Schaffner A, Jelalian E, Hart CN, Scholl TO, Munoz-Christian K, Yin E, Phipps MG, Keadle S, Abrams B. Randomized controlled clinical trial of behavioral lifestyle intervention with partial meal replacement to reduce excessive gestational weight gain. Am J Clin Nutr. 2018 Feb 1;107(2):183-194. doi: 10.1093/ajcn/nqx043. PMID 29529157
- [Derived] Clifton RG, Evans M, Cahill AG, Franks PW, Gallagher D, Phelan S, Pomeroy J, Redman LM, Van Horn L; LIFE-Moms Research Group. Design of lifestyle intervention trials to prevent excessive gestational weight gain in women with overweight or obesity. Obesity (Silver Spring). 2016 Feb;24(2):305-13. doi: 10.1002/oby.21330. Epub 2015 Dec 26. PMID 26708836

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: Participants in the enhanced-usual care group received all aspects of usual care offered by their prenatal care providers, including physicians, nurses, nutritionists, or counselors from the Women, Infants, and Children's Special Supplemental Nutrition Program (WIC)
Period: Overall Study
Arm/Group | Standard Care | Lifestyle Intervention
Started | 132 | 132
Completed | 127 | 129
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who withdrew (N = 7) are not included in baseline analysis population table or in any results.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Lifestyle Intervention | Total
Number analyzed (Participants) | 128 | 129 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (5.5) | 30.7 (5.3) | 30.3 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 129 | 257
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 53 | 107
  Not Hispanic or Latino | 74 | 76 | 150
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 128 | 129 | 257

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain Per Week of Observation
Description: Rate of gestational weight gain will be computed as difference between weights measured at study entry and gestational week 35; this difference will be divided by the number of weeks of observation during pregnancy (i.e., weeks between study entry and final pregnancy assessment). If gestational week 35 is unavailable, most proximal clinic visit weight will be used.
Time Frame: 13 weeks gestation, 35 weeks gestation
Measure: Least Squares Mean (Standard Deviation); unit: kg/wk
Arm/Group | Standard Care | Lifestyle Intervention
Number analyzed (Participants) | 127 | 129
kg/wk | 0.39 (0.23) | 0.33 (0.25)

2. Secondary Outcome: Offspring Weight Gain
Description: Offspring weight for age z scores from birth (1 week), to 6 months, and 12 months of age.
Time Frame: 1 week, 6 months, 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Kcals/Day
Description: Changes in maternal calorie intake (Kcal/day)
Time Frame: 13 weeks gestation, 34 weeks gestation
Measure: Least Squares Mean (95% Confidence Interval); unit: kcals/day
Arm/Group | Standard Care | Lifestyle Intervention
Number analyzed (Participants) | 128 | 129
kcals/day
  13 weeks | 1777 [1681 to 1873] | 1743 [1649 to 1837]
  34 weeks | 1785 [1685 to 1888] | 1673 [1570 to 1776]

4. Secondary Outcome: Changes in Offspring Dietary Intake
Description: Changes in offspring intake of breast milk (#feeds per day) and/or formula (#feeds per day).
Time Frame: 1 week, 6 months, 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Maternal Glucose
Description: Fasting glucose
Time Frame: 13 weeks gestation, 34 weeks gestation
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Standard Care | Lifestyle Intervention
Number analyzed (Participants) | 127 | 129
mg/dL
  13 weeks | 84 [84 to 88] | 87 [85 to 88]
  34 weeks | 85 [83 to 86] | 83 [81 to 84]

6. Secondary Outcome: Number of Women Exceeding IOM Guidelines as a Proportion of Total Number of Women in Each Group.
Description: Self-reported pre-pregnancy weight will be subtracted from weight measured at last clinic visit prior to delivery. Women will be categorized as exceeding 2009 IOM guidelines if the difference is > 11.5 kg gain for women with prepregnancy overweight or >9 kg for women with prepregnancy obesity.
Time Frame: 13 weeks, 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Lifestyle Intervention
Number analyzed (Participants) | 127 | 129
Participants | 69 | 53

7. Secondary Outcome: Number of Women at or Below Prepregnancy Weight as a Proportion of the Total Number of Participants in Each Group
Description: Weight measured at 48-56 weeks postpartum and subtracted from self-reported prepregnancy weight and then categorized as at or below vs. above self-reported prepregnancy weight.
Time Frame: 48-56 weeks post delivery
Measure: Count of Participants; unit: Participants
Groups:
- Standard Care: Participants in the enhanced-usual care group received all aspects of usual care offered by their prenatal care providers, including physicians, nurses, nutritionists, or counselors from the Women, Infants, and Children's Special Supplemental Nutrition Program (WIC) (
Arm/Group | Standard Care | Lifestyle Intervention
Number analyzed (Participants) | 128 | 129
Participants | 38 | 41

ADVERSE EVENTS:
Time Frame: 35 weeks gestation
Description: Preterm delivery (< 36 weeks)
Arm/Group | Standard Care | Lifestyle Intervention
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/129
Other Adverse Events (participants affected / at risk) | 5/128 | 4/129
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=128) | Lifestyle Intervention (N=129)
Preterm Delivery (General disorders) | 5 (5) | 4 (4) — <36 weeks gestation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No